CLINICAL TRIAL: NCT04048200
Title: The Effect of Opioid Free Anesthesia on the Postoperative Opioid Consumption in Laparoscopic Bariatric Surgeries: Randomized Controlled Study
Brief Title: The Effect of Opioid Free Anesthesia in Bariatric Surgeries
Acronym: Opioidfree
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 33107/05/19; Tanta University (Other: Faculty of Medicine, Tanta University)
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Adverse Effect of Drugs and Medicaments in Therapeutic Use; Adverse Effects in the Therapeutic Use of Anaesthetics
Keywords: Dexmedetomidine; Ketamine; Fentanyl; Bariatric surgeries
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Intervention Model Description: Prospective study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinded study Closed sealed envelops will be used to make the participants blind to their group.
  The continuous infusion regimen in the syringe pump will be prepared by anesthesia resident who will not participating in the the study . It will contain normal saline in control group and actual dexmedetomidine and ketamine in the other group. This will make the investigator blind to the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Anesthesia will be induced by fentanyl 1 ug/kg, propofol 2 mg/kg, and rocuronium 1 mg/kg to facilitate tracheal intubation. After endotracheal intubation, the patients will be connected to mechanical ventilator with its parameters adjusted to maint5ain etCO2 32-36 mmhg. Anesthesia will be maintained by sevoflurane 2% in a mixture of oxygen: Air 1: 1 to maintain entropy 40-60. The patients in this group will be connected to a syringe pump before induction of anesthesia that was prepared by anesthesia resident not participating in the study and contain normal saline and adjusted at a rate of 1 ml/kg/hr till the end of the surgery.
  Interventions: Drug: Fentanyl
- Opioid free anesthesia group (Experimental): A syringe 50 ml was prepared by anesthesia resident not participating in the study and contain 100 ug of dexmedetomidine (2 ug/ml) and 25 mg ketamine 90.5 mg/ml) and 200 mg lidocaine (4 mg/ml). The syringe will be connected to the patients before induction of anesthesia at a rate of 0.1 ml/kg/hr according to the ideal body weight. Anesthesia will be induced by propofol 2 mg/kg, and rocuronium 1 mg/kg to facilitate tracheal intubation. After endotracheal intubation, the patients will be connected to mechanical ventilator with its parameters adjusted to maint5ain etCO2 32-36 mmhg. Anesthesia will be maintained by sevoflurane 2% in a mixture of oxygen: Air 1: 1 to maintain entropy 40-60. The syringe infusion will be continued till the end of peritoneal manipulation. Patients in this group will receive magnesium sulphate preload at a dose of 40 mg/kg ideal body weight followed by maintenance infusion of 10 mg/kg/hr.
  Interventions: Drug: Dexmedetomidine Ketamine

INTERVENTIONS:
Drug: Fentanyl — Anesthesia will be induced by fentanyl, propofol, and rocuronium with maintenance of anesthesia using sevoflurane.
  Other Names: Opioid based Anesthesia
  Arms: Control group
Drug: Dexmedetomidine Ketamine — No opioid will be used in induction of anesthesia. A combination of dexmedetomidine and ketamine will be infused. Sevoflurane will be used for maintenance of anesthesia.
  Other Names: Opioid sparing
  Arms: Opioid free anesthesia group

SUMMARY:
This is a prospective randomized controlled study that will be carried out on morbid obese patients admitted to Tanta University hospitals for laparoscopic bariatric surgeries. The patients will be randomly assigned into;- Control group:- Anesthesia will be induced by fentanyl 1 ug/kg, propofol 2 mg/kg, and rocuronium 1 mg/kg to facilitate tracheal intubation. Anesthesia will be maintained by sevoflurane 2% in a mixture of oxygen: Air 1: 1 to maintain entropy 40-60.

Opioid free anesthesia group;- Anesthesia will be induced by propofol 2 mg/kg, rocuronium 1 mg/kg to facilitate tracheal intubation. After endotracheal intubation, and a combination of dexmedetomidine and ketamine infusion. Anesthesia will be maintained by sevoflurane 2% in a mixture of oxygen: Air 1: 1 and continuing the infusion of dexmedetomidine and ketamine o maintain entropy 40-60.

DETAILED DESCRIPTION:
This prospective randomized controlled study will be carried out on patients who will be presented for laparoscopic bariatric surgery in the general surgery department in Tanta university hospitals over six-month duration that will start immediately after obtaining ethical committee approval and clinical trial registration. An informed written consent will be obtained from all the participants, all patients data will be confidential and will be used for the current study only.

Inclusion criteria:

Morbid obese patients with BMI 40-50 kg/m2 aged more than 21 years and American Society of Anesthesiologists Class III presented for laparoscopic sleeve gastrectomy or gastric bypass.

Exclusion criteria:

* Patients refused to participate.
* Patients with known or suspected or known allergy to the used medication.
* Patients with moderate to severe obstructive sleep apnea
* Patients with uncontrolled blood sugar, cardiac, renal, or hepatic functions.
* Patients receiving opioids preoperatively
* Uncooperative patients
* Patients received preoperative gabapentoids.

Anesthetic technique Once the patients will arrive to the operating room, intravascular access will be established, fluid preload will be started, and basic monitor will be attached.

The patients will be randomly distributed into two equal groups by the aid of computer-generated software of randomization: - ▪ Control group (30 patients): Anesthesia will be induced by fentanyl 1 ug/kg, propofol 2 mg/kg, and rocuronium 1 mg/kg to facilitate tracheal intubation. After endotracheal intubation, Anesthesia will be maintained by sevoflurane 2% in a mixture of oxygen: Air 1: 1 to maintain entropy 40-60. The patients in this group will be connected to a syringe pump before induction of anesthesia that was prepared by anesthesia resident not participating in the study and contain normal saline and adjusted at a rate of 1 ml/kg/hr till the end of the surgery.

▪ Opioid free anesthesia group (30 patients): A syringe 50 ml was prepared by anesthesia resident not participating in the study and contain 100 ug of dexmedetomidine (2 ug/ml) and 25 mg ketamine 90.5 mg/ml) and 200 mg lidocaine (4 mg/ml). The syringe will be connected to the patients before induction of anesthesia at a rate of 0.1 ml/kg/hr according to the ideal body weight. Anesthesia will be induced by propofol 2 mg/kg, and rocuronium 1 mg/kg to facilitate tracheal intubation. Anesthesia will be maintained by sevoflurane 2% in a mixture of oxygen: Air 1: 1 to maintain entropy 40-60. The syringe infusion will be continued till the end of peritoneal manipulation. Patients in this group will receive magnesium sulphate preload at a dose of 40 mg/kg ideal body weight followed by maintenance infusion of 10 mg/kg/hr.

In both groups, routine anti-emetic prophylaxis will be administrated composed of ondansetron 4 mg and dexamethasone 8 mg before the surgery. Additional analgesia will be provided using 1 gm of paracetamol together with intraperitoneal local anesthetics and wound infiltration.

All the patients will be connected to the bispectral index monitor with maintaining its value 40-60. Increase in n bispectral index value above 60 will be managed by additional dose of fentanyl 0.5 ug/kg IBW and increasing the concentration of sevoflurane by 0.2% till the value decreased below 60.

At the end of the surgery, the inhalational anesthesia will be switched off with reversal of muscle relaxation using neostigmine and atropine with full awake extubation of the patient. The patients will be transported to the recovery room for adequate postoperative monitoring and management.

Measurements:

1. Patient age, weight, height.
2. The total dose consumption of fentanyl consumed intraopeartively.
3. The total volume consumed of sevoflureane intraoperatively (ml/hr).
4. The postoperative Visual Analogue Score (VAS): It will be measured every 2 hours till 6 h, then every 4 h till 24 h. In case of increase the VAS more than 3, a rescue analgesia will be administrated in the form of 2mg morphine i.v that may be repeated.
5. The time for the first request of morphine rescue analgesia
6. The total dose of morphine consumed in the first 24 h after surgery
7. The recovery profile of the patient.
8. Patients satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obese patients with BMI 40-50 kg/m2
* Aged more than 21 years and American Society of Anesthesiologists Class III
* Presented for laparoscopic sleeve gastrectomy or gastric bypass.

Exclusion Criteria:

* Patients refused to participate.
* Patients with known or suspected or known allergy to the used medication.
* Patients with moderate to severe obstructive sleep apnea
* Patients with uncontrolled blood sugar, cardiac, renal, or hepatic functions.
* Patients receiving opioids preoperatively
* Uncooperative patients
* Patients received preoperative gabapentoids.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | The first 24 hours postoperatively
  The total dose of morphine consumed postoperative as a rescue analgesia to maintain the VAS less than 4

SECONDARY OUTCOMES:
Intraoperative sevoflurane consumption | Through out the whole intraoperative period
  The intraoperative consumption of sevoflurane in ml per one hour

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Ismaiel, M.D, Principal Investigator — Lecturer of Anesthesia and Intensive Care, Tanta University
Locations (1):
- Tanta University hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
Once the study had been successfully completed, the data will be shared for other researchers.